CLINICAL TRIAL: NCT00960323
Title: A One-Directional, Open-Label Drug Interaction Study to Investigate the Effects of Multiple-Dose Atorvastatin on the Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Colchicine and Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1019
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — Colchicine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine Alone (Active Comparator): baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Atorvastatin (Experimental): Colchicine pharmacokinetics in the presence of atorvastatin at steady state.
  Interventions: Drug: Atorvastatin; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone in the morning on Day 1.
  Arms: Colchicine Alone
Drug: Atorvastatin — Atorvastatin (1 x 40 mg tablet) administered once daily on Days 15-28.
  Arms: Colchicine with Atorvastatin
Drug: Colchicine — A single dose of 0.6 mg colchicine administered with a single dose of 40 mg atorvastatin in the morning on Day 28 after an overnight fast.
  Arms: Colchicine with Atorvastatin

SUMMARY:
Colchicine is a substrate for cytochrome P450 3A4 (CYP3A4). In-vitro studies have indicated that the ortho-and para-hydroxylated metabolites of atorvastatin may be CYP3A4/5 competitive and mechanism-based inhibitors (MBI). This study will evaluate the effect of multiple doses of atorvastatin on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Colchicine is a substrate for cytochrome P450 3A4 (CYP3A4). In-vitro studies have indicated that the ortho-and para-hydroxylated metabolites of atorvastatin may be CYP3A4 /5 competitive and mechanism-based inhibitors (MBI). This study will evaluate the effect of multiple doses of atorvastatin on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. Twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of colchicine (1 x 0.6 mg tablet) on Day 1 after an overnight fast. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose at times sufficient to adequately define the pharmacokinetics of colchicine. After a 14 day washout period, starting on the morning of Day 15 and continuing through Day 27, subjects will return to the clinic for once daily administration of atorvastatin (1 x 40 mg tablet) after an overnight fast. After taking the first dose of atorvastatin on Day 15, subjects will remain in the clinic for 1 hour post-dose administration for observation. On the morning of Day 28 after an overnight fast, all study participants will receive a co-administered single oral dose of colchicine (1 x 0.6 mg tablet) and atorvastatin (1 x 40 mg tablet). Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose at times sufficient to adequately define the pharmacokinetics of colchicine in the presence of atorvastatin at steady state. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse, respiratory rate and temperature will be measured at screening, baseline and upon study discharge. Blood pressure and pulse will also be measured pre-dose and at 1 and 2 hours post-dose on Days 1 and 28 to coincide with peak plasma concentrations of colchicine and atorvastatin. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive
* Hemoglobin greater than or equal to 11.5g/dL

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine or atorvastatin or any other HMG-CoA reductase inhibitor agents (i.e. simvastatin, lovastatin, rosuvastatin, fluvastatin, and pravastatin)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Davis MW, Wason S. Effect of steady-state atorvastatin on the pharmacokinetics of a single dose of colchicine in healthy adults under fasted conditions. Clin Drug Investig. 2014 Apr;34(4):259-67. doi: 10.1007/s40261-013-0168-8. PMID 24452746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-two volunteers were screened for participation in this study. Eight were screen failures, four were not needed, four withdrew consent and two had a schedule conflict.
Groups:
- Colchicine, Atorvastatin, Colchicine and Atorvastatin: On the morning of Day 1, subjects received a single dose of colchicine 0.6 mg after an overnight fast, followed by a 14 day washout period. On the mornings of Days 15-27, subjects received a daily dose of atorvastatin 40 mg after an overnight fast. On the morning of Day 28, subjects received a co-administered single oral dose of colchicine 0.6 mg and atorvastatin 40 mg following an overnight fast.
Period: Colchicine Alone
Arm/Group | Colchicine, Atorvastatin, Colchicine and Atorvastatin
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine, Atorvastatin, Colchicine and Atorvastatin
Started | 24
Completed | 24
Not Completed | 0
Period: Atorvastatin Alone
Arm/Group | Colchicine, Atorvastatin, Colchicine and Atorvastatin
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Colchicine and Atorvastatin
Arm/Group | Colchicine, Atorvastatin, Colchicine and Atorvastatin
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine, Atorvastatin, Colchicine and Atorvastatin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.29 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Colchicine
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing on Days 1 and 28 and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hours after dose administration.
Population: 24 subjects were enrolled in this study. One subject withdrew from the study prior to Period II check in due to a schedule conflict.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: On the morning of Day 1, subjects received a single dose of colchicine 0.6 mg after an overnight fast followed by a 14 day washout period.
- Colchicine With Atorvastatin: On the morning of Day 28, subjects received a co-administered single oral dose of colchicine 0.6 mg and atorvastatin 40 mg after an overnight fast.
Arm/Group | Colchicine Alone | Colchicine With Atorvastatin
Number analyzed (Participants) | 23 | 23
pg/mL | 2,023.29 (903.14) | 2,487.96 (646.99)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule for colchicine.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Groups:
- Colchicine Alone: On the morning of Day 1, subjects received a single dose of colchicine 0.6 mg after an overnight fast, followed by a 14 day washout period.
Arm/Group | Colchicine Alone | Colchicine With Atorvastatin
Number analyzed (Participants) | 23 | 23
pg*hr/mL | 8,717.33 (4,208.19) | 10,714.92 (4,060.71)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. [AUC(0-∞)] was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant for colchicine.
Time Frame: as for outcome 1
Population: 24 subjects were enrolled in this study. One subject withdrew prior to Period II check-in. The pharmacokinetic parameter, AUC(0-∞), could not be determined for 1 subject in the Colchicine Alone group and for 4 subjects in the Colchicine with Atorvastatin group.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Colchicine Alone | Colchicine With Atorvastatin
Number analyzed (Participants) | 22 | 19
pg*hr/mL | 9,592.53 (3,349.19) | 11,043.58 (3,867.03)

ADVERSE EVENTS:
Description: 24 subjects were enrolled in this study. One subject withdrew consent prior to Period II check-in.
Groups:
- Atorvastatin Alone: On the mornings of Days 15-27, subjects received a daily dose of atorvastatin 40 mg after an overnight fast.
- Colchicine and Atorvastatin: On the morning of Day 28, subjects received a co-administered single oral dose of colchicine 0.6 mg and atorvastatin 40 mg after an overnight fast.
Arm/Group | Colchicine Alone | Atorvastatin Alone | Colchicine and Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 4/24 | 6/24 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Alone (N=24) | Atorvastatin Alone (N=24) | Colchicine and Atorvastatin (N=23)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days